CLINICAL TRIAL: NCT03115502
Title: Hemodynamic Changes and Vascular Tone Control After Bariatric Surgery. Prognostic Value Regarding Hypertension and Target Organ Damage
Brief Title: Hemodynamic Changes and Vascular Tone Control After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Anna Oliveras, Head of Hypertension & Vascular Risk Unit. Nephrology Department, Parc de Salut Mar
Other Study IDs: Baritha
Record Dates: First submitted 2016-01-13; First posted 2017-04-14 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Systemic Vascular Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Obese patients have increased cardiovascular risk and target organ damage (TOD) as compared to people with normal weight. Weight loss reduces cardiovascular risk and TOD. These changes have been associated mainly to changes in inflammatory and pro-atherogenic markers. Office peripheral blood pressure (BP) appears to decrease after bariatric surgery, but information on changes in 24h-ambulatory-BP-monitoring (24h-ABPM) and central-BP(cBP), or about the possible role of renin-angiotensin-aldosterone (RAAS), serotonin(STS) and endocannabinoid(ECS) systems is scarce. Our hypothesis is that the hemodynamic changes mediated by alterations in the RAAS, STS and ECS after weight loss are also responsible for the reduction of TOD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 - 65 years,
2. who have medical indication for treatment with bariatric surgery and agreeing to undergo the intervention,with
3. given informed consent

Exclusion Criteria:

1. Unmeeting the above Inclusion Criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 - 65 years, who have medical indication for treatment with bariatric surgery and agreeing to undergo the intervention.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-08; Primary Completion 2018-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Mean changes 24h-aortic systolic-blood pressure (SBP) measured in mmHg | From baseline to the final exam (12 months) with intermediate evaluations at 1, 3 and 6 months.

SECONDARY OUTCOMES:
Mean changes in aortic- 24h, daytime and nighttime blood pressure estimates others than 24h systolic blood pressure measured in mmHg | From baseline to the final exam (12 months) with intermediate evaluations at 1, 3 and 6 months.
Mean changes in peripheral- 24h, daytime and nighttime blood pressure estimates measured in mmHg | From baseline to the final exam (12 months) with intermediate evaluations at 1, 3 and 6 months.
Mean change in office blood pressure estimates measured in mmHg | From baseline to the final exam (12 months) with intermediate evaluations at 1, 3 and 6 months.
Mean change in arterial stiffness parameters (I) | From baseline to the final exam (12 months) with intermediate evaluations at 1, 3 and 6 months.
  pulse wave velocity measured in m/s
Mean change in arterial stiffness parameters (II) | From baseline to the final exam (12 months) with intermediate evaluations at 1, 3 and 6 months.
  augmentation index measured in %
Mean change in Left ventricular mass index | From baseline to the final exam (12 months) with intermediate evaluations at 1, 3 and 6 months.
  Left ventricular mass index measured in g/m2
Mean change in Left atrium diameter | From baseline to the final exam (12 months) with intermediate evaluations at 1, 3 and 6 months.
  Left atrium diameter measured in mm
Mean change in Ejection fraction | From baseline to the final exam (12 months) with intermediate evaluations at 1, 3 and 6 months.
  Ejection fraction measured in %,
Mean change in left ventricular remodeling index | From baseline to the final exam (12 months) with intermediate evaluations at 1, 3 and 6 months.
  left ventricular remodeling index, do not have units
Mean change in carotid intima-media thickness measured in mm | From baseline to the final exam (12 months) with intermediate evaluations at 1, 3 and 6 months.
Mean change in biochemical parameters measured in mg/dl or mmol/L | From baseline to the final exam (12 months) with intermediate evaluations at 1, 3 and 6 months.
Mean change in the components of the renin-angiotensin system | From baseline to the final exam (12 months) with intermediate evaluations at 1, 3 and 6 months.
  renin-angiotensin system: plasma renin activity: ng/mL/h, plasma aldosterone: pg/ml, angiotensinogen: mng/100ml, angiotensin 1-7: pg/ml, ACE: UI/l, ACE-2: UI/I
Mean change in the serotonergic system components | From baseline to the final exam (12 months) with intermediate evaluations at 1, 3 and 6 months.
  serotonergic system: 5-HIAA:ng/ml, 5-HT:ng/mL
Mean change in the components of the endocannabinoid system | From baseline to the final exam (12 months) with intermediate evaluations at 1, 3 and 6 months.
  endocannabinoid system: Anandamide: nmol/mL, 2-arachidonoylglycerol: mg/ml
Mean change in pro-atherosclerotic markers | From baseline to the final exam (12 months) with intermediate evaluations at 1, 3 and 6 months.
  pro-atherosclerotic markers: omentine-1: ng/ml, chemerine: ng/ml, leptin: ng/ml, adiponectine: mcg/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar_Nefrology, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oliveras A, Molina L, Goday A, Sans L, Riera M, Vazquez S, Benaiges D, Granados AM, Ramon JM, Pascual J. Effect of bariatric surgery on cardiac structure and function in obese patients: Role of the renin-angiotensin system. J Clin Hypertens (Greenwich). 2021 Jan;23(1):181-192. doi: 10.1111/jch.14129. Epub 2020 Dec 17. PMID 33331692
- [Derived] Oliveras A, Goday A, Sans L, Arias CE, Vazquez S, Benaiges D, Ramon JM, Pascual J. Changes in Central 24-h Ambulatory Blood Pressure and Hemodynamics 12 Months After Bariatric Surgery: the BARIHTA Study. Obes Surg. 2020 Jan;30(1):195-205. doi: 10.1007/s11695-019-04107-9. PMID 31346932